CLINICAL TRIAL: NCT02364869
Title: Effect of Prebiotic (Fructooligosaccharide) on Uremic Toxins and Cardiovascular Markers of Chronic Kidney Disease Patients
Brief Title: Prebiotic in Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Universidade Federal do Paraná (Other); Pontifícia Universidade Católica do Paraná (Other)
Responsible Party: Principal Investigator, Lilian Cuppari, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCTI/CNPQ: 449614/2014-0
Record Dates: First submitted 2015-01-13; First posted 2015-02-18 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Disease
Keywords: P-cresyl sulfate; Indoxyl sulfate; Intestine; Endothelial function
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — fructooligosaccharide; Prebiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fructooligosaccharide (Experimental): 12g daily, for 12 weeks
  Interventions: Dietary Supplement: Fructooligosaccharide
- Maltodextrin (Placebo Comparator): 12g daily, for 12 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Fructooligosaccharide — Patients will be evaluated at baseline, week 6 and 12.
  Other Names: Prebiotic
  Arms: Fructooligosaccharide
Dietary Supplement: Maltodextrin — Placebo Comparator. Patients will be evaluated at baseline, week 6 and 12.
  Arms: Maltodextrin

SUMMARY:
This 12-week double-blind randomized controlled clinical trial aims to investigate the effect of a prebiotic (fructooligosaccharide - FOS) on serum and urinary levels of uremic toxins (p-cresyl sulfate and indoxyl sulfate) of non-dialysis dependent CKD patients, and the impact of such intervention on cardiovascular markers, intestinal permeability, endotoxemia and inflammatory response.

DETAILED DESCRIPTION:
Intestinal microbiome has been considered a new therapeutic target for chronic kidney disease (CKD) due to its potential role on the metabolic disturbances associated to the disease. The abnormalities in the microbiota, frequently found in patients with CKD, contribute to the accumulation of uremic toxins derived from the unbalanced fermentation of nitrogen compounds in relation to the non-digestible carbohydrates. Among them, p-cresyl sulfate and indoxyl sulfate have been associated with inflammation, kidney disease progression, endothelial dysfunction and increased risk of death in this population. Preliminary studies especially on hemodialysis have shown that the use of prebiotic, probiotic and symbiotic may represent a promising intervention due to their beneficial effect as modulators of the intestinal microbiota that might promote a reduction on serum concentration of p-cresyl sulfate and indoxyl sulfate. In comparison to probiotic, prebiotic have the advantage to stimulate the host's microbiota and to occur naturally in several foods. In the context of CKD, the use of prebiotics has been poorly investigated. Therefore, the primary aim of this study is to investigate the effect of a prebiotic (fructooligosaccharide - FOS) on serum and urinary levels of p-cresyl sulfate and indoxyl sulfate of non-dialysis dependent CKD patients. As a secondary aim we will investigate the impact of such intervention on cardiovascular markers, intestinal permeability, endotoxemia and inflammatory response. This is a 12-week double-blind randomized controlled clinical trial. Fifty non-diabetic patients with CKD stages 3a and 4 will be randomly assigned to a 12 g/day of FOS or maltodextrin (placebo). The serum and urinary concentrations of p-cresyl sulfate and indoxyl sulfate will be determined by high performance liquid chromatography (HPLC). The assessment of endothelial function includes ultrasonography of the brachial artery, measurement of plasma and urinary nitric oxide, monocyte chemoattractant protein 1 (MCP1), stromal cell-derived factor 1 alpha (SDF1α), oxide - trimethylamine N- (TMAO), ambulatory blood pressure monitoring (ABPM) and pulse wave velocity (PWV). The serum intestinal trophic markers (glucagon-like peptide 2 - GLP2 - and epidermal growth factor - EGF), intestinal permeability (Zonulin), endotoxemia and inflammation (IL-6 and CRP) will be determined by ELISA. Food intake will be assessed by 3-day food records. Protein intake will be estimated by calculating the protein equivalent of nitrogen appearance (PNA). The Bristol Scale, the Roma III Criteria and the Gastrointestinal Symptoms Rating Scale will be applied to evaluate gastrointestinal effects during the follow-up. The subjective global assessment questionnaire, the spectroscopic bioimpedance analysis and the handgrip strength will be applied to evaluate the nutritional status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years
* Estimated glomerular filtration rate between 45 to 15 ml/min/1,73m².

Exclusion Criteria:

* diabetes mellitus, malignance, severe liver disease, autoimmune diseases, congestive heart failure class III / IV, HIV, history of gastrointestinal disease
* use of phosphate binders, laxatives or prebiotic, probiotic, symbiotic, antibiotics, immunosuppressants and / or anti-inflammatory drugs three months preceding the study.
* patients using laxatives who refuse to stop treatment during the follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Uremic toxicity evaluated by serum and urinary levels of p-cresyl sulfate and indoxyl sulfate | 12 weeks

SECONDARY OUTCOMES:
Endotoxemia measured by serum levels of lipopolysaccharides | 12 weeks
Intestinal permeability evaluated by serum levels of Zonulin | 12 weeks
Intestinal epithelium evaluated by serum levels of glucagon-like peptide 2 (GLP2) | 12 weeks
Intestinal epithelium evaluated by serum levels of epidermal growth factor (EGF). | 12 weeks
Inflammation measured by serum levels of Interleukin-6 (IL-6) | 12 weeks
Inflammation measured by serum levels of c-reactive protein (CRP) | 12 weeks
Endothelial function evaluated by ultrasonography of the brachial artery | 12 weeks
Endothelial function evaluated by blood pressure monitoring (ABPM) | 12 weeks
Endothelial function evaluated by pulse wave velocity (PWV). | 12 weeks
Endothelial function evaluated by plasma and urinary levels of nitric oxide | 12 weeks
Endothelial function evaluated by plasma and urinary levels of monocyte chemoattractant protein 1 (MCP1) | 12 weeks
Endothelial function evaluated by plasma and urinary levels of stromal cell-derived factor 1 alpha (SDF1α) | 12 weeks
Endothelial function evaluated by plasma and urinary levels of oxide - trimethylamine N- (TMAO) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Cupari, PhD, Principal Investigator — Affiliate professor of Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148